CLINICAL TRIAL: NCT04370379
Title: A Dose Escalation Phase I Clinical Study to Evaluate the Tolerability and Safety of IBI302 in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Trial to Evaluate the Safety and Tolerability of Repeated Intravitreal Injection of IBI302 in Neovascular AMD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI302A102
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — IBI302; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose of IBI302 (Experimental)
  Interventions: Drug: IBI302 (the first dose level)
- high dose of IBI302 (Experimental)
  Interventions: Drug: IBI302 (the second dose level)
- 2mg aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: IBI302 (the first dose level) — q4week (3 injections) followed by PRN dosing
  Arms: low dose of IBI302
Drug: IBI302 (the second dose level) — q4week (3 injections) followed by PRN dosing
  Arms: high dose of IBI302
Drug: Aflibercept — 2mg, q4week (3 injections) followed by q8week
  Arms: 2mg aflibercept

SUMMARY:
This study is designed for multi-center, open-label, randomized, dose escalation phase I trial to evaluate the safety and tolerability of a multiple dose intravitreal injection of IBI302 in neovascular AMD patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria

1. Male or female patient ≥ 50 yrs. of age.
2. Active subfoveal or parafoveal CNV secondary to neovascular AMD.
3. Willing and able to sign informed consent form and comply with visit and study procedures per protocol.

Exclusion criteria

1. Presence of uncontrolled glaucoma in the study eye (defined as IOP≥30mmHg despite the standardized treatment);
2. Presence of active intraocular or periocular inflammation or infection;
3. History of severe hypersensitivity/allergy to active ingredients or any excipients of the study drug, or fluorescein and povidone iodine;
4. Participated in any clinical study of any other drug within three months prior to enrollment, or attempted to participate in other drug trials during the study;
5. Diabetic patients have any of the following conditions:HbA1c>7.5% when screening;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Ocular safety, assessed by BCVA, slitlamp examination, ophthalmoscopy, IOP, fundus photography | Baseline to Day140
Incidence of adverse events | Baseline to Day140

SECONDARY OUTCOMES:
Changes in central subfield thickness by OCT compared with baseline | Baseline to Day140
Changes in CNV characteristics and CNV area by FA compared with baseline | Baseline to Day140
Changes in BCVA compared with baseline | Baseline to Day140
Positive rate of anti-drug antibody and neutralizing antibody of IBI302 | Baseline to Day140
the area under the drug-time curve from 0 to time t of IBI302 | Baseline to Day140
the area under the curve at the time of 0-infinity of IBI302 | Baseline to Day140
The peak concentration of IBI302 | Baseline to Day140
The peak time of IBI302 | Baseline to Day140
Clearance rate of IBI302 | Baseline to Day140
Half-life of IBI302 | Baseline to Day140
VEGF concentration | Baseline to Day140
Concentration of complement fragments | Baseline to Day140

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jia H, Li T, Sun J, Gong Y, Liu H, Wang H, Chen J, Liu W, Lu S, Feng L, Wan Q, Qian L, Wang F, Liu X, Sun X. A Novel Bispecific Fusion Protein Targeting C3b/C4b and VEGF in Patients With nAMD: A Randomized, Open-Label, Phase 1b Study. Am J Ophthalmol. 2023 Apr;248:8-15. doi: 10.1016/j.ajo.2022.11.016. Epub 2022 Nov 21. PMID 36410472